CLINICAL TRIAL: NCT00758173
Title: A Population Based Study of Genetic Predisposition and Gene-Environment Interactions in Prostate Cancer in East Anglia, Trent and West Midlands
Brief Title: Study of Genes and the Environment in Patients With Prostate Cancer Residing in the East Anglia, Trent, or West Midlands Regions of the United Kingdom
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cancer Research UK (Other)
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: CDR0000589199; MREC-SEARCH-PROSTATE
Record Dates: First submitted 2008-09-22; First posted 2008-09-23 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2008-09

CONDITIONS: Prostate Cancer
Keywords: prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Amplified Fragment Length Polymorphism Analysis

INTERVENTIONS:
Genetic: polymorphism analysis
Other: laboratory biomarker analysis
Other: questionnaire administration

SUMMARY:
RATIONALE: Studying samples of blood from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This study is looking at genetic susceptibility and the interactions between genes and the environment in patients with prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To obtain epidemiological information and biological material on a population-based series of prostate cancer cases.
* To identify novel cancer susceptibility genes by comparison of genotype frequencies in cases with the corresponding frequencies in large control series.
* To estimate the age and sex-specific risks associated with variants in predisposition genes.
* To evaluate interactions between polymorphisms in predisposition genes and potential lifestyle risk factors.

OUTLINE: This is a multicenter study.

Patients complete a detailed epidemiological questionnaire, including information on education, occupation, smoking habits, alcohol consumption, height, weight, family history of cancer, and past medical history.

Blood samples are collected from patients. DNA is extracted from these blood samples and from samples collected from cancer-free control participants in MREC-SEARCH-CONTROL as well as from additional controls through the European Prospective Investigation of Cancer (EPIC) study (a population based study of diet and health based in Norfolk, East Anglia). DNA samples are analyzed for polymorphisms of low penetrance cancer susceptibility genes.

In addition to the prostate cancer patients recruited for this study, patients with breast, ovarian, endometrial, colorectal, bladder, kidney, pancreatic, brain and esophageal cancer, malignant melanoma, and lymphoma cancer are recruited in the following related clinical trials: MREC-SEARCH-BREAST, MREC-SEARCH-OVARIAN, MREC-SEARCH-ENDOMETRIAL, MREC-SEARCH-COLORECTAL, and MREC-SEARCH-CANCER.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of prostate cancer within the past 5 years
* Identified through the cancer registry serving any of the following geographic regions of the United Kingdom:

  * East Anglia
  * Trent
  * West Midlands

PATIENT CHARACTERISTICS:

* Identified by the patient's general practitioner as fit to contact for this study
* No serious mental illness or retardation

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 18 Years to 74 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2008-02

PRIMARY OUTCOMES:
Acquisition of epidemiological information and biological material
Identification of novel cancer susceptibility genes
Estimation of the age and sex-specific risks associated with variants in predisposition genes
Evaluation interactions between polymorphisms in predisposition genes and potential lifestyle risk factors

CONTACTS AND LOCATIONS:
Overall Officials: Paul Pharoah, MD, Study Chair — Cancer Research UK
Locations (1):
- University of Cambridge Cancer Research UK, Cambridge, England, United Kingdom